CLINICAL TRIAL: NCT02894827
Title: The Effect of When Medication is Taken on Nutritional Status in Hospitalized Patients Older Than 65 Years
Acronym: MEDICANUT2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VAN WYMELBEKE 2015
Record Dates: First submitted 2016-08-31; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Nutritional Status
MeSH Terms: interventions — Blood Specimen Collection; Flow Cytometry; Blotting, Western

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- EMS
  Interventions: Biological: Blood sample; Other: Flow cytometry; Other: western blot
- Control
  Interventions: Biological: Blood sample; Other: Flow cytometry; Other: western blot

INTERVENTIONS:
Biological: Blood sample
Other: Flow cytometry
Other: western blot

SUMMARY:
Polypathology in elderly subjects requires polypharmacy but even though the efficacy of a medication and digestive tolerance are ensured, the medication can be taken a long time from meals to reduce its side-effects. Despite numerous studies that have investigated links between medication and malnutrition, none have assessed the influence of the time the drug is taken on the evolution of the nutritional status of elderly hospitalized persons. So as to identify the best nutritional criterion in hospitalized persons, a retrospective pilot study will be conducted in about thirty patients. Their medication will be recorded and their nutritional status will be evaluated using the Geriatric Nutritional Risk Index (GNRI), albumin, prealbumin levels, weight and the Mini Nutritional Assessment (MNA) short form.

This preliminary study will allow us to choose the best nutritional criterion to compare the impact of two strategies for taking medication (post prandial versus pre-prandial) on improving the nutritional status of malnourished elderly hospitalized patients taking multiple drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years or more.
* patients with a stable or controlled acute disease hospitalized in a geriatric follow-up care unit.
* patients whose life expectancy is greater than 30 days.
* patients able to eat food normally.
* patients able to swallow their medication.
* patients with at least 3 drugs to be taken orally per day, not including oral nutritional supplements.

Exclusion Criteria:

* patients at the end of life.
* patients whose drugs must be taken before meals like Non-steroid anti-inflammatory drugs (NSAIDs), glinides, oral antidiabetic agents (OAD).
* patients with parenteral and/or enteral nutrition in the period preceding admission to the geriatric unit.
* patients with indications for parental and/or enteral nutrition.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients with a stable or controlled acute disease hospitalized in a geriatric follow-up care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
MNA short form | 30 days

SECONDARY OUTCOMES:
Geriatric Nutritional risk form | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France